CLINICAL TRIAL: NCT02686645
Title: Fecal Microbiota Therapy for Recurrent Clostridium Difficile Infection
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Ian Davis, Assistant Professor Department of Medicine, Dalhousie University, Queen Elizabeth II Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSHA REB File #: 1020563
Record Dates: First submitted 2016-01-25; First posted 2016-02-19 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Clostridium Difficile Infection
Keywords: Fecal Microbiota Transplantation
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation; Vancomycin; Loperamide; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fecal Microbiota Therapy (Experimental): Vancomycin 125 mg po qid for 7 days or metronidazole 500 mg po tid for 7 days pre-treatment. Loperamide 4 mg po after morning prep and 2 mg post treatment. The route of administration fecal microbiota will be by retention enema via a rectal tube.
  Interventions: Biological: Fecal Microbiota; Drug: vancomycin; Drug: Loperamide; Drug: metronidazole

INTERVENTIONS:
Biological: Fecal Microbiota — The fecal microbiota will be by retention enema administered through a rectal tube.
Drug: vancomycin — All subjects will be pre-treated with vancomycin 125 mg po qid X 7 days prior to the fecal microbiota.
Drug: Loperamide — The subject will take 4 mg of loperamide after the morning bowel prep (approximately 1 hour prior to the procedure) and 2 mg again after the procedure.
Drug: metronidazole — If unable to tolerate vancomycin, then it will be substituted with metronidazole 500 mg po tid X 7 days prior to the fecal microbiota.

SUMMARY:
Interventional, single arm, single-centre trial to evaluate the effectiveness and safety of fecal microbiota therapy (FMT) in the investigators population.

DETAILED DESCRIPTION:
This is a study of the effects of FMT for the treatment of patients with recurrent Clostridium difficile infection (CDI). The investigators plan to enrol approximately 5-10 patients per year over the next 5 years to a maximum of 50 patients. Patients with recurrent CDI referred to the designated Gastrointestinal (GI) or Infectious Diseases (ID) services will be screened for inclusion and exclusion by the primary investigator (PI), sub investigators and/or designated study personnel.

Those patients meeting the criteria will be offered FMT and will be the recipient. An informed consent will be obtained from both the recipient and the donor prior to proceeding with the study protocol. Demographic information as well as details of the medical history and results of standard laboratory tests will be collected on the recipients and donors.

The donor preferably should be < 60 years old to maximize the fecal microbiota. As this does involve biological samples there is a theoretical risk of transmission of an infectious agent. To minimize this risk, the donors will be selected preferentially from a spouse or sexual partner. If this is not possible, then another relative or acquaintance would serve as the donor as identified by the recipient. In either case, the donor will be screened for potentially transmissible infections. This will include a health screening questionnaire adapted from Canadian Blood Services, a clinical examination and laboratory investigations to rule out known transmissible infectious diseases. The donor will complete a satisfaction survey.

The submitted stool will be processed in the lab as per the "Stool Prep Protocol". The route of administration will be by retention enema via a rectal tube. As the treatment is not an emergency the investigators will have the option, if necessary, to store the stool for future treatment. If the sample is not used it will be discarded at 90 days and another sample will be obtained if still required.

Prior to the treatment the recipient will also submit a sample of stool. Along with this a portion of the donor sample will be stored in at -80 degrees C for future molecular tests to determine the diversity of the microbiota. This may be performed at a later date dependent on obtaining the necessary funding.

Recipients will be followed for 6 months post FMT to monitor for success of treatment, adverse reactions, recipient satisfaction and a quality of life assessment.

note: if laboratory testing for Clostridium difficile (CD) changes the new test will replace the cytotoxicity test.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥ 18 yrs of age.
2. Recurrent CDI despite two courses of standard treatment (ie. 10 days of oral vancomycin or metronidazole) and a 6 week taper of oral vancomycin.
3. Laboratory confirmation of CDI by enzyme immunoassay (EIA), cytotoxicity assay and/or polymerase chain reaction (PCR).
4. Presence of persistent diarrhea defined as ≥ 3 loose or watery bowel movements in 24hr continuing for >2 days and diarrhea ongoing at the time of inclusion.

Exclusion Criteria:

1. Severely immunosuppressed patients will not be enrolled. This is defined as >20 mg prednisone/d for >1 month, recent transplant patients (haematological <2yrs and solid organ < 6 months), transplant with active graft versus host disease, HIV (with CD4<200), immunosuppressive antibody treatment (eg. tumour necrosis factor inhibitor, rituximab), other high dose long term systemic immunosuppression) and severe congenital immunodeficiency.
2. Age <18 years old.
3. Pregnancy.
4. Patient expected to expire in < 30d.
5. Current hospital admission for an indication other than CDI or need for vasopressor medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Resolution of CDI | 30 days
  Resolution of CDI will be defined as < 3 bowel movements per day for 7 consecutive days or stool negative for Clostridium difficile (CD) on 2 consecutive stool sample at least 1 day apart within 30 days of the treatment.

SECONDARY OUTCOMES:
Success of treatment | 3 months
  Success of treatment with be absence of recurrence of CDI within 3 months of treatment. A recurrence will be defined as ≥ 3 bowel movements per day after a period of resolution with a positive stool for CD toxin within 3 months for treatment.
Adverse effects | 6 months
  Adverse effects experienced with treatment up to 6 months after treatment.
Quality of life | day 0, 3 months and 6 months
  Quality of Life Assessment (prior to, 3 month and 6 months after FMT) using the Short Form 36 (SF-36) Health Survey.
Recipient Satisfaction | 1week, 3 months and 6 months
  Recipient Satisfaction Survey which will be completed within 1 week of the FMT and again at 3 and 6 months post FMT.
Donor Satisfaction | 1 week
  The donor will complete a satisfaction survey within 1 week after the stool donation.

CONTACTS AND LOCATIONS:
Overall Officials: Ian R Davis, MD,FRCPC, Principal Investigator — Dalhousie University, Department of Medicine, Division Infectious Diseases

IPD SHARING:
Plan to Share IPD: No